CLINICAL TRIAL: NCT02500225
Title: Ulku Ozgul, Associate Professor, Inonu University, Department of Anesthesiology and Reanimation
Brief Title: Comparison the Effects of Etomidate and Sevoflurane During Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Associate Professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Ulku 1
Record Dates: First submitted 2015-07-09; First posted 2015-07-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; ECT
Keywords: Etomidate; Sevoflurane
MeSH Terms: interventions — Etomidate; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etomidate (Active Comparator): 0.2 mg/kg etomidate during anesthesia induction
  Interventions: Drug: Etomidate; Drug: Sevoflurane
- 8% sevoflurane (Active Comparator): Sevoflurane 8% concentration during anesthesia induction
  Interventions: Drug: Etomidate; Drug: Sevoflurane

INTERVENTIONS:
Drug: Etomidate — 0.2 mg/kg etomidate
  Other Names: Hypnomidate
Drug: Sevoflurane — 8% Sevoflurane
  Other Names: Sevorane

SUMMARY:
The purpose of the study was to investigate the effects of etomidate or sevoflurane used in electroconvulsive therapy (ECT) on duration of seizure, hemodynamic response and recovery profiles.

DETAILED DESCRIPTION:
Twenty-five patients will be a total of 150 ECT treatments in this prospective, double-blinded, crossover study. Each patient will receive either 0.2 mg/kg etomidate (Group 1) or 8% sevoflurane (Group 2) in 100% oxygen at 6 L/min fresh gas flow until loss of consciousness for their initial electroconvulsive therapy session. In subsequent sessions, patients will receive the alternative sevoflurane concentration and then alternated between doses until the sixth session. Muscle paralysis will achieve with 1 mg/kg succinylcholine. Motor (EMG) and electroencephalography seizure duration (EEG), heart rate (HR) and mean arterial pressure (MAP) values, and recovery times will recorde.

ELIGIBILITY:
Inclusion Criteria:

* Study include 25 patients of American Society of Anesthesiologists (ASA) physical status I-II aged between 18-60 years who schedule for ECT sessions under general anesthesia

Exclusion Criteria:

* Pregnancy
* Cerebrovascular disease
* Epilepsy
* Unstable cardiovascular disease
* Chronic obstructive pulmonary disease; and
* Renal or hepatic failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Motor (EMG) seizure duration | intraoperative
  Motor seizure duration in electroconvulsive therapy
electroencephalography (EEG) seizure duration | intraoperative
  seizure duration in electroconvulsive therapy

SECONDARY OUTCOMES:
heart rate (HR), | (approximately 5 minutes for all measurements) prior to the seizure, after the anesthetic induction, and following the ECT session at 1 minute, 3 minutes, and 10 minutes
  heart rate in electroconvulsive therapy
mean arterial pressure (MAP) | (approximately 5 minutes for all measurements) prior to the seizure, after the anesthetic induction, and following the ECT session at 1 minute, 3 minutes, and 10 minutes
  MAP will be measured by a blood pressure cuff
recovery times | (approximately 5 minutes for all measurements) prior to the seizure, after the anesthetic induction, and following the ECT session at 1 minute, 3 minutes, and 10 minutes
  Recovery times will be assessed with spontaneous breathing, eye opening, obeying commands times

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, MD, Study Director — Inonu University School of Medicine

REFERENCES:
- [Result] Janouschek H, Nickl-Jockschat T, Haeck M, Gillmann B, Grozinger M. Comparison of methohexital and etomidate as anesthetic agents for electroconvulsive therapy in affective and psychotic disorders. J Psychiatr Res. 2013 May;47(5):686-93. doi: 10.1016/j.jpsychires.2012.12.019. Epub 2013 Feb 9. PMID 23399487
- [Result] Toprak HI, Gedik E, Begec Z, Ozturk E, Kaya B, Ersoy MO. Sevoflurane as an alternative anaesthetic for electroconvulsive therapy. J ECT. 2005 Jun;21(2):108-10. doi: 10.1097/01.yct.0000166633.73555.28. PMID 15905753